CLINICAL TRIAL: NCT05418569
Title: The Impact of a Locally Tailored Evidence-based Chinese Smartphone Application in Management of Type 1 Diabetes Mellitus Aged 6-18 Years in Hong Kong - a Randomized Controlled Trial
Brief Title: Chinese Smartphone App for 6-18 Years With T1DM - RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEE LAI KA SAMANTHA, Honorary Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PR-HKCH-13
Record Dates: First submitted 2022-05-29; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Type1 Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm - Use of the new smartphone application for T1DM (Active Comparator): The use of the locally designed smartphone application for T1DM for 6 months, which contained the following domains:
  * Type 1 DM self-management information and decision-making algorithm
  * Carbohydrate counting information on local food in Hong Kong
  * DM day-to-day troubleshooting psychosocial scenarios
  * Game-based interactive tools for DM knowledge enhancement
  * Usage tracking for each domain of the smartphone application
  * Individual participant identification and access code (known to research assistant)
  Interventions: Device: Intervention arm - A new smartphone application for pediatric type 1 DM
- Control Arm - Standard diabetic education (Placebo Comparator): Received standard diabetic care (diabetic nurse education and regular follow-ups) with optional use of an existing smartphone application for general diabetic information for both adult and pediatric population (that encompasses both information for type 1 and type 2 DM)
  Interventions: Other: Standard diabetic eduction

INTERVENTIONS:
Device: Intervention arm - A new smartphone application for pediatric type 1 DM — An evidence-based locally tailored Chinese smartphone application for pediatric type 1 DM
  Arms: Intervention Arm - Use of the new smartphone application for T1DM
Other: Standard diabetic eduction — Received standard diabetic care (diabetic nurse education and regular follow-ups) with optional use of an existing smartphone application for general diabetic
  Arms: Control Arm - Standard diabetic education

SUMMARY:
Moving into the era of electronic communication, it changes the way we shall engage our children and adolescents. According to data of the Census and Statistics Department of Hong Kong releases in 2019, more than 80% and up to 99.4% of those aged 10-14 years, and aged 15-24 years respectively had a mobile phone device. A recent survey carried by Kebede et al. (2019) had shown that using diabetes apps was positively associated with self-care behavior in type 1 and type 2 diabetes mellitus (DM). A systematic review carried in Spain by Quevedo Rodríguez et al. (2018) had found most of the available smartphone apps lacked quality certification and very few provide scientific references on their content.

In Hong Kong, there is currently no Chinese smartphone application targeting for the pediatric type 1 population, therefore, most of the education is based on face-to-face or telephone communication with the diabetic nurse and endocrinologists in limited encounters. For families or patients with limited command of English language, apart from one adult oriented DM information smartphone application, the chance of having on-hand mobile device support is truly limited. In light of this context, we shall first design an evidence-based locally tailored Chinese smartphone application for pediatric type 1 DM and then evaluate its effectiveness in improving management of type 1 DM in a robust manner.

The main research question for this project is whether a self-help smartphone application in local Chinese language, tailored to include local clinical practice, culture and food spectrum, can improve diabetes control and psychological wellbeing in patients with type 1 diabetes mellitus aged 6-18 years. Eligible participants will be randomized to either using the smartphone application (on top of standard diabetic care) or continue standard diabetic care. The study aims to compare the difference between the two groups for their diabetic control and the psychological wellbeing.

DETAILED DESCRIPTION:
Objectives To evaluate the impact of a locally designed evidence-based Chinese smartphone application in improving type 1 diabetes mellitus management for aged 6-18 years in Hong Kong.

Hypothesis Use of smartphone application can improve diabetes mellitus control and self-care ability, psychological wellbeing and quality of life.

Design and subjects A single-blinded randomized controlled trial employing block randomization. Inclusion criteria: (1) Type 1 diabetes mellitus diagnosed for at least 6 months, (2) Aged 6-18 years, (3) HbA1c >/=6.0%, (4) Receiving DM care in Hong Kong. Exclusion criteria: (1) Lack of the ability to use a smartphone application, (2) Moderate to severe visual impairment, (3) Cannot read Chinese language. Aim for 57 participants in each of the control and intervention arms for a statistical power of 80%.

Study instruments

(1) HemoglobinA1c, (2) Time in range and frequency of hypoglycaemia by continuous glucose monitoring, (3) Chinese versions of PSC-35, PedsQL and DSMQ questionnaires.

Interventions Use of the smartphone application for 6 months.

Main outcome measures Primary outcomes include (1) HbA1c, (2) Time in range, (2) Frequency of hypoglycaemia. Secondary outcomes are scores of PSC-35, PedsQL and DSMQ.

Data analysis and expected results Data to be analysed with intention-to-treat. A post hoc analysis is planned to capture data in the reduced application usage group. Generalized estimating equation will be employed to analyse the data involving within-subject covariance. Around 10% dropout rate assumed. A statistically significant result is defined by a 2-tailed alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Known type 1 DM diagnosed for at least 6 months
2. Aged 6-18 years
3. HbA1c >/= 6.0% in the preceding 6 months prior to recruitment
4. Receiving DM care in Hong Kong

Exclusion Criteria:

1. Lack of the ability to use a smartphone application despite an introduction session the smartphone application intended for this study
2. Moderate to severe visual impairment that may affect the smartphone application usage
3. Cannot read Chinese language.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months (Assessed at 3 months and 6 months from start of intervention)
  A decrease of 0.5% is considered significant
CGM data | 6 months
  Time in range, glycemic variability and percentage of hypoglycemia as documented by continuous glucose monitoring (for a period of 2 weeks) at baseline and at the end of study.
Self/Parent-reported questionnaires on hypoglycemia frequency | 6 months
  Self/Parent-reported questionnaires on hypoglycemia frequency, the lowest glucose reading during hypoglycemia and number of severe hypoglycemia requiring glucagon use - to be performed at baseline and at the end of study.

SECONDARY OUTCOMES:
The PSC-35 (Pediatric Symptom Checklist-35 items) questionnaires | 6 months
  The PSC-35 (Pediatric Symptom Checklist-35 items) questionnaires is employed to assess the psychological wellbeing at baseline and at the end of study.
The Chinese version of the Diabetes Self-Management Questionnaire (DSMQ) | 6 months
  The Chinese version of the Diabetes Self-Management Questionnaire (DSMQ) is employed to assess the diabetes self-management behavior at baseline and at the end of study. The data on the questionnaire's use in youths or children are not available yet. We will interpret with caution for those questions not entirely applicable to participants <18 years.
The Chinese version of the Pediatric Quality of Life Inventory 4.0 plus the 3.0 diabetes module | 6 months
  The Chinese version of the Pediatric Quality of Life Inventory 4.0 plus the 3.0 diabetes module to be filled in at baseline and at the end of study.Diabetes module will not be required for participants with ages 5-7 years as Chinese version is currently not available.
Self/Parent-reported questionnaires to assess on carbohydrate counting accuracy on local Hong Kong diet at baseline and at the end of study | 6 months
  Self/Parent-reported questionnaires to assess on carbohydrate counting accuracy on local Hong Kong diet at baseline and at the end of study
Self-reported smartphone application usage satisfaction | 6 months
  Self-reported smartphone application usage satisfaction to be filled at 3 months and the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Samathan Lee, Principal Investigator — Hong Kong Children's Hospital
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong